CLINICAL TRIAL: NCT04226170
Title: A Phase II, Study to Evaluate the Safety and Tolerability of Pyridostigmine When Given With Ondansetron to Subjects With Anti-AchR Positive Myasthenia Gravis
Brief Title: Study of Pyridostigmine With Ondansetron in Subjects With Anti-AchR Positive Myasthenia Gravis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: DAS-MG, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS-001-001
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-05

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: randomized to ondansetron + pyridostigmine or placebo+ pyridostigmine in a 3:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only unblinded study member will be the pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment (Active Comparator): ondansetron + pyridostigmine
  Interventions: Drug: DAS-001
- Placebo (Placebo Comparator): placebo+ pyridostigmine
  Interventions: Drug: DAS-001

INTERVENTIONS:
Drug: DAS-001 — ondansetron + pyridostigmine

SUMMARY:
This is a phase II, single center, randomized, double-blind, placebo-controlled, study in patients with a diagnosis of anti-AchR antibody positive myasthenia gravis.

DETAILED DESCRIPTION:
Methodology: This is a phase II, randomized, double-blind, placebo-controlled, study in patients with a diagnosis of anti-AchR antibody positive myasthenia gravis.

Study Design: The clinical trial will be conducted over a 6-week treatment period with 2 groups.

* Group A: Patients currently taking pyridostigmine and experiencing pyridostigmine-related gastrointestinal (GI) adverse events (AEs) within the past 14 days.
* Group B: Patients not currently taking pyridostigmine due to a documented history of GI AEs.

Randomized to either the control (pyridostigmine+ placebo) or the test group (pyridostigmine + ondansetron) and treated for 6 weeks. Following enrolment, patients may (if needed) titrate up their pyridostigmine dose at the investigator's discretion each week to the highest dose deemed appropriate, tolerable and safe.

ELIGIBILITY:
Inclusion criteria

1. Male and female subjects aged 18 years old and up who have been diagnosed with anti-AchR antibody positive myasthenia gravis.
2. Subjects can be either:

   currently taking pyridostigmine and after Lead-in Period experience dose limiting GI AEs related to pyridostigmine (must include nausea, vomiting or diarrhea) during Lead-in
3. Subjects must be willing and able to complete a GI symptom diary within a consistent timeframe on a daily basis.
4. Must be clinically stable in judgement of treating neurologists for past 3 months.
5. Must be positive for acetylcholine receptor antibodies.
6. Subjects must be able to swallow liquid.
7. Subjects must be in otherwise good health as determined by their medical history, physical examination, vital signs, and laboratory tests. A subject with a medical abnormality may be included only if the investigator or designee considers that the abnormality will not introduce significant additional risk to the subject's health or interfere with study objectives.
8. Subjects must have signed an informed consent form indicating that they understand the purpose of, and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions.

Exclusion criteria:

1. Any acute or chronic diseases which are associated with GI distress (such as nausea, vomiting, or diarrhea), which could interfere with the subjects' safety during the trial, expose them to undue risk, or interfere with the study objectives.
2. History or presence of hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
3. History of substance abuse, known drug addiction, or positive test for drugs of abuse or alcohol.
4. Patients currently using marijuana for any reason (medical or recreational).
5. Known hypersensitivity to pyridostigmine, or to ondansetron or similar 5-HT3 serotonin receptor antagonists.
6. ECG changes including QT interval prolongation and congenital long QT syndrome. Electrolyte abnormalities (e.g., hypokalemia or hypomagnesemia), congestive heart failure, bradyarrhythmia's or other medicinal products that lead to QT prolongation.
7. Treatment with drugs affecting peripheral cholinergic transmission within 1 month of study entry (with the exception of pyridostigmine).
8. Subjects unlikely to co-operate during the study, and/or be questionably compliant in the opinion of the investigator.
9. Patients currently being treated with narcotics.
10. Patients being treated with aminoglycoside antibiotics, which are contraindicated in myasthenia gravis.
11. Patients unable to be contacted in case of an emergency.
12. Intake of an investigational drug within 30 days of study entry.
13. Pregnancy and women of childbearing potential not willing to follow the birth control requirements as described in the informed consent or breastfeeding.
14. History or presence of obstructive pulmonary disease or urinary obstruction (contraindication for pyridostigmine).
15. This use of selective serotonin reuptake inhibitors (SSRIs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with change in the gastrointestinal (GI) side effects | 6 weeks
  difference in GI side effects as measured by the GSRS-self (Gastrointestinal System Rating Scale - self-administered)

SECONDARY OUTCOMES:
Number of participants with change in the side effects | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" . Incidence and nature of adverse events
Number of participants with change in in physical examine | 6 weeks
  physical examination changes General appearance,Head, eyes, ears, nose, and throat, Respiratory, Cardiovascular, Musculoskeletal, Abdomen, Neurologic, Extremities, Dermatologic, Lymphatic)
Number of participants with change in in clinical laboratory evaluations | 6 weeks
  changes in clinical laboratory evaluations (Creatinine, Potassium(K+),Sodium (Na+) , Chloride (Cl-), Magnesium (Mg++), Calcium, Inorganic phosphate, Glucose, Urea,Bilirubin (Total) ,Bilirubin (direct), AST, ALT, GGT, Alkaline phosphatase, Total Protein, Albumin,Hematocrit Hemoglobin Platelet count Red blood cell (RBC) count WBC count WBC differential Mean cell volume (MCV) Mean cell hemoglobin (MCH) MCH concentration (MCHC)
Number of participants with change in Electrocardiography (ECG) | 6 weeks
  ECG (standard digital 12-lead in singlicate)
Plasma concentrations of pyridostigmine | 6 weeks
  Cmax
Plasma concentrations of ondansetron | 6 weeks
  Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No